CLINICAL TRIAL: NCT00288366
Title: Anticonvulsant Mood Stabilizers, Antipsychotic Drugs and the Insulin Resistance Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Alliance for Research on Schizophrenia and Depression (Other); Pfizer (Industry)
Responsible Party: Principal Investigator, Herbert Meltzer, Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 050942; NARSAD
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Results first posted 2019-08-06 (Actual); Last update posted 2019-08-06 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder
Keywords: schizophrenia; schizoaffective disorder; bipolar disorder; metabolic syndrome
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): aripiprazole (Abilify)
  Interventions: Drug: ziprasidone vs. aripiprazole; Drug: aripiprazole vs. ziprasidone
- 2 (Active Comparator): ziprasidone (Geodon)
  Interventions: Drug: aripiprazole vs. ziprasidone

INTERVENTIONS:
Drug: ziprasidone vs. aripiprazole — ziprasidone vs. aripiprazole dosed according to package insert
  Arms: 1
Drug: aripiprazole vs. ziprasidone — aripiprazole vs. ziprasidone dosed according to package insert

SUMMARY:
The objective of this study is to determine the effect of various mood stabilizers (MS) on the insulin resistance syndrome (IRS; also called the metabolic syndrome) alone and in patients treated with antipsychotic drugs (APDs). Patients will be switched from their current antipsychotic medication to aripiprazole (Abilify) or ziprasidone (Geodon) (unless clinically contraindicated) for comparison with metabolic levels during treatment with the former medication.

The metabolic syndrome is an empirical concept based on extensive evidence that a constellation of 5 metabolic abnormalities, e.g. increased cholesterol, hypertension, low HDL, taken together, predict marked increases in the risk of CVD, stroke and some types of cancer.

ELIGIBILITY:
Inclusion criteria

To be eligible, patients must :

* Be male or female, age 18-65
* Be diagnosed with schizophrenia, schizoaffective disorder or bipolar disorder with psychotic features according to DSM-IV criteria
* Be currently receiving antipsychotic drugs (clozapine, haloperidol, olanzapine, quetiapine, or risperidone) (APDs) alone, mood stabilizer(s) (MS) alone, or a combination of the two
* Have a history of compliance with the above medication
* Have presumptive IRS as indicated by a TG/HDL ratio > 3.5 on current antipsychotic medication
* Be Medicaid eligible or maintain insurance covering requested lab procedures
* Be able to provide written informed consent Exclusion criteria

A patient will be considered ineligible if he/she:

* Has a diagnosis other than schizophrenia, schizoaffective disorder or bipolar disorder with psychotic features according to DSM-IV criteria.
* Has a history of noncompliance with prescribed psychiatric medications
* Has a TG/HDL ratio < 3.5 on current medication
* Is uninsured or is unable to self-pay potential costs of required lab procedures not covered by insurance.
* Is unable to provide written informed consent.
* (Females only) Is pregnant, lactating or plans to become pregnant during study participation

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2006-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yuejin Chen, M.D., Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Psychiatric Hospital at Vanderbilt, Nashville, Tennessee, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Aripiprazole: aripiprazole (Abilify)
  ziprasidone vs. aripiprazole: ziprasidone vs. aripiprazole dosed according to package insert
  aripiprazole vs. ziprasidone: aripiprazole vs. ziprasidone dosed according to package insert
- Ziprasidone: ziprasidone (Geodon)
  aripiprazole vs. ziprasidone: aripiprazole vs. ziprasidone dosed according to package insert
Period: Overall Study
Arm/Group | Aripiprazole | Ziprasidone
Started | 23 | 26
Completed | 23 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Aripiprazole | Ziprasidone | Total
Number analyzed (Participants) | 23 | 26 | 49
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 23 | 26 | 49
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (8.5) | 45.5 (9.4) | 44.9 (8.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 16 | 29
  Male | 10 | 10 | 20
Region of Enrollment [Number; unit: participants]
  United States | 23 | 26 | 49

OUTCOME MEASURES:

1. Primary Outcome: HDL Ratio
Description: change in HDL ratio after medication switch
Time Frame: 24 weeks from Baseline
Measure: Mean (Standard Error); unit: unit of Measure ''g/dL''
Arm/Group | Aripiprazole | Ziprasidone
Number analyzed (Participants) | 23 | 26
unit of Measure ''g/dL''
  Baseline | 39.7 (1.6) | 38.4 (1.5)
  24 weeks | 43.5 (2.1) | 42.3 (1.8)

ADVERSE EVENTS:
Arm/Group | Aripiprazole | Ziprasidone
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/26
Other Adverse Events (participants affected / at risk) | 1/23 | 0/26
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Aripiprazole (N=23) | Ziprasidone (N=26)
Worsening of psychiatric symptoms (Nervous system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes